CLINICAL TRIAL: NCT05605353
Title: Exploiting the Gut Microbiota and Its Metabolites in Pelvic Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-066-22
Record Dates: First submitted 2022-10-20; First posted 2022-11-04 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Neoplasm
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will undertake 16srRNA gene sequencing of the bacterial DNA, metabolite and Short Chain fatty acid analysis from the blood and faecal samples (taken from the right colon at the time of the operation). Comparisons between these microbial analysis will then be undertaken in a pair-wise approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Colorectal: Patients with rectal or colon cancer
  Interventions: Diagnostic Test: Faecal microbiota sampling and blood sampling
- Gynaecological: Patients with uterine, ovarian or cervical cancers
  Interventions: Diagnostic Test: Faecal microbiota sampling and blood sampling
- Urological: Patients with bladder or prostate cancers
  Interventions: Diagnostic Test: Faecal microbiota sampling and blood sampling

INTERVENTIONS:
Diagnostic Test: Faecal microbiota sampling and blood sampling — There is no intervention in this study. We will obtain faeces and blood from the recruited patients and assess the microbiota and their metabolites therein. This is an observational work

SUMMARY:
The large intestine is the last part of the digestive tract. It absorbs water and dietary substances. However, it is also where most of our bacteria are resident. These bacteria are important for our health and influence many different diseases, including Colon Cancer, Ulcerative Colitis and Crohn's disease. The gut bacteria can also potentially influence responses to treatments in other cancers by helping to change the responses to radiotherapy and chemotherapy. The interactions between these bacteria and the rest of our cells are only now becoming understood and there is little research on the interactions between these bacteria and cancer radiotherapy treatments in pelvic cancer.

We will therefore explore this in more detail. We will ask for samples of the patient's poo before their treatment for pelvic cancers. This will include patients with bladder, prostate, cervical, ovarian, womb or colorectal cancers. By doing so we will be able to compare the profile of gut bacteria with responses to treatments, thereby increasing our understanding of the colonic bacteria.

To do this we process the poo specimens to remove the bacterial genetic material (DNA) of the bacteria and process it on a machine to read the genetic code and also study the metabolites that they will produce. We can then make a direct comparison between different samples of the relative numbers of different bacteria present. In some cases, we will compare this to metabolites and inflammatory and immune markers identified in a blood sample. This work might help future patients by determining what are the best bacteria to have in the colon during cancer treatments. These could potentially be given to patients, before their cancer treatment, in the form of probiotic medications, should there be an improvement demonstrated in our research. Alternatively we could alter the patients' intakes of specific dietary fibres to boost these bacteria specifically.

DETAILED DESCRIPTION:
The University of Aberdeen and Aberdeen Royal Infirmary (ARI) in NHS Grampian are in the unique position of having a single site campus for microbiota-related laboratory science at the world-famous Rowett Institute, Biorepository facilities on campus for rapid sample processing and NHS facilities for treatment of multiple pelvic tumour types, including colorectal, gynaecological and urological.

Patients will be approached in their respective pelvic cancer clinics, after identification for potential inclusion at the respective multi-disciplinary team (MDT) meeting. The patient will be informed of their diagnosis and management plan by a clinician responsible for their care (may include Clinical Nurse Specialist). Patients will only be approached about the research at a subsequent meeting, e.g. when the specialist nurses contact the patient to address any further questions around the management plan discussed, they attend the consultant clinic for consent to definitive treatment, etc. This gives the patient sufficient time to process their diagnosis and management plan before introducing the research. At this meeting patients will be provided with the PIS (this will be posted to the patient if the meeting is via video teleconference). If they are willing to consider being involved, they will then be contacted by a research nurse or other suitably qualified team member, who will discuss the study further and answer any questions. If they are willing to take part arrangements will be made for a member of the clinical team to obtain written informed consent when the patient attends hospital for a subsequent clinical appointment.

They will be asked to donate a faecal sample (and in a subset of colorectal patients, a right-sided colonic contents sample taken at the time of their operation) for processing at the Rowett Institute Human Nutrition Unit before the start of their next cancer therapy (chemotherapy, radiotherapy or surgery). Consent will also be sought to obtain a blood sample. This will normally be obtained during routine venesection for clinical reasons and will be blood surplus to clinical requirements processed by the Biorepository. Where necessary, if blood is not being collected as part of standard clinical care, an extra venepuncture, of 5mls, will be requested. Blood will be processed for plasma extraction.

Patients will also be encouraged to complete an optional food frequency questionnaire (FFQ) indicating what they have eaten and drank in the three months before taking their stool samples. However, if they feel unable to complete this, their decision will be respected and they can continue in the study. These questionnaires take around 30 minutes to complete and will be provided to the patients either during a clinical appointment before their first cancer therapy or posted out to them. A subgroup of patients will also be asked if they would be willing to provide a more in-depth assessment of their diet on the four days before providing the stool sample but it will be highlighted to them that this is optional and they are free to refuse.

Faecal samples will be collected from the ARI brought to the hospital on the day of a clinic appointment or initial treatment for the patient. Alternatively, the participant can leave the sample at a specific drop off centre in the Rowett institute. This will be left to the discretion of the participant as to whichever is most convenient for them. Completed food diaries/questionnaires will also be collected at the same time and in the same location as the faecal sample drop-off.

No other additional samples are required from the patient. After obtaining the specimens, at the Rowett Institute, a portion will be processed by Dispomix for DNA extraction using Powersoil DNA extraction kits and stored in freezers before analysis by 16S rRNA gene sequencing. Another portion will be processed and stored for SCFA analysis by gas chromatography and some of the remaining faeces stored for future analyses.

Plasma will be extracted from the blood samples from the NHS Haematology laboratories and transferred to the Rowett Institute by the research team involved in the study. In situations where a blood sample has not been taken for clinical purposes the blood sample will be collected by a phlebotomist or other trained staff at the Human Nutrition unit of the Rowett Institute. Once the plasma has been extracted, the blood samples will be stored in freezers at the Rowett Institute.

16S rRNA gene sequencing of faecal DNA will be undertaken at the Centre for Genome Enabled Biology and Medicine (CCEBM), University of Aberdeen, including bioinformatics analysis. Using 16S rRNA gene sequencing, a small portion of the bacterial genetic material is examined, which differs between different bacteria, allowing us to estimate the 'relative abundance' of each within each specimen. We will also analyse SCFAs in faeces by GC and plasma by GC-MS (this more sensitive technique is required for plasma due to lower concentrations of metabolites present) at the Rowett Institute Analytical facility. At the end of this study, if sufficient sample remains in a usable condition we would like to store this for future research. After necessary funding and approvals are obtained we may in future investigate bacterial DNA in more detail (to species/strain level) by metagenomics and other metabolites, e.g. tryptophan, bile acids, and inflammatory (e.g. calprotectin) and immune markers (e.g. cytokines).

Clinical data will be pseudo-anonymised at source and collected by the research team (including biobank staff for baseline data and, research nurses, clinical fellows, radiographers, etc, for follow up data). This will be included in the subsequent analysis. Tumour responses and the side effects of radiotherapy/ chemoradiotherapy or surgery will be obtained from patient notes to look at toxicity and outcomes, and some patients will have been asked to fill in questionnaires as part of their routine clinical follow-up, such as the RTOG and EPIC26 (questionnaires routinely used in clinical practice).

16S rRNA gene sequencing data will be analysed by Bioinformaticians at the University of Aberdeen specialised in handling these large data sets, to determine the richness and relative abundance of bacteria present. Data will be stored by IT services on the High Performance Computer Cluster and submitted to a public repository. Associations will be studied between 16S rRNA gene sequencing data, SCFA analysis and available clinical data. Statistical analysis will be undertaken by Statisticians from Biomathematics and Statistics Scotland

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to consent
2. Any patient who is being treated in NHS Grampian for a pelvic cancer (Colorectal, urological or gynaecological) above 16 years of age

Exclusion Criteria:

1. patients who are not willing to consent to be involved
2. Malignancies from other sources or anatomical locations
3. Patients who lack the understanding of the study to obtain appropriate levels of consen

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 450 patients who have been diagnosed with pelvic neoplasms in the NHS Grampian region of Scotland, United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between microbial analysis and response to cancer therapy | 18 month recruitment
  To assess if key microbes (analysed by pyrosequencing), or their metabolic byproducts (analysed by short chain fatty acid identification) detect for positive or adverse response to conventional therapy and cancer outcomes

SECONDARY OUTCOMES:
Are there differences in the gut microbiota between urological, colorectal and gynaecological cancers? | 18 month recruitment
  16srRNA pyrosequencing and short chain fatty acid analysis will be undertaken for patients with the three cancer groupings. These data will be compared against each other to assess similarity or differences in the faecal microbial flora between the conditions.

CONTACTS AND LOCATIONS:
Overall Officials: George Ramsay, FRCS, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be pseudo-anonymised at source and held strictly within the principles of the UK GDPR legislation. Thus, individual participant data will not be available to other researchers.